CLINICAL TRIAL: NCT04099537
Title: Evaluating the Effect of Approach Avoidance Training on Action Tendencies for Individuals With Skin Picking Disorder
Brief Title: Skin Picking Approach Avoidance Task
Acronym: SPAAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Milwaukee (Other)
Responsible Party: Principal Investigator, Han Joo Lee, Professor, University of Wisconsin, Milwaukee
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPAAT2018
Record Dates: First submitted 2019-03-09; First posted 2019-09-23 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Skin-Picking
Keywords: skin picking; cognitive training; approach-avoidance
MeSH Terms: conditions — Excoriation Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Approach cognitive training (Experimental): This training is a single session training. Each session lasts about 30 minutes where participants are to pull the joystick toward (approach) them when seeing skin stimuli on a computer screen.
  Interventions: Behavioral: Computerized cognitive training
- Avoidance cognitive training (Experimental): This training is a single session training. Each session lasts about 30 minutes where participants are to push the joystick away (avoidance) from them when seeing skin stimuli on a computer screen.
  Interventions: Behavioral: Computerized cognitive training
- Placebo cognitive training (Placebo Comparator): This training is a single session training. Each session lasts about 30 minutes where participants are to push and pull the joystick towards or away from them (no rule) when seeing skin stimuli on a computer screen.
  Interventions: Behavioral: Computerized cognitive training

INTERVENTIONS:
Behavioral: Computerized cognitive training — Participants are trained to approach or avoid stimuli of skin using a joystick. Participants are to pull or push the joystick toward or away when skin stimuli are present. Thus, behaviorally, there may be an increase, decrease, or no change in approach tendencies towards skin.

SUMMARY:
Pathological skin picking (PSP) is conceptualized as a behavioral addiction. Research has shown that behavioral addictions (e.g., problematic alcoholism or smoking) can be reduced using a cognitive retraining tool called approach-avoidance training (AAT). Participants will be randomly assigned to a single-session of AAT: (a) approach training, (b) avoidance training, or (c) placebo training and will be assessed at baseline, post-training (i.e., 30 minutes after training), and 2-week follow up. The investigators hypothesize that those in the approach training will show greater reduction in approach tendencies at post-treatment and 2-week follow up, compared to those in the approach training or placebo conditions. This study may produce data that will guide the development of a training program that focuses on the maladaptive action tendencies in skin picking symptoms.

DETAILED DESCRIPTION:
Pathological Skin Picking (PSP) is one of many debilitating Body Focused Repetitive Behaviors (BFRBs) that involves repetitive picking to gain the gratification of relieving anxiety or tension. Thus, this behavior may cause infections, lesions, and scarring, resulting in psychosocial impairment or medical attention. Because of the habitual/compulsive nature of the disorder, researchers conceptualize this maladaptive coping mechanism as a behavioral addiction which may occur without conscious awareness. Therefore, it is important to identify the automatic motivational orientations behind BFRBs. There is compelling evidence to suggest that a novel technological behavior paradigm, called Approach Avoidance Training (AAT), can be used to assess and modify action tendencies (i.e., approach or avoidance) in behavioral addictions like PSP. This game-like task has the participant push (=avoid) or pull (=approach) a joystick based on a target and control stimulus presented on a computer screen. This push-pull paradigm is in response to the individual's inherent action tendencies.

The overarching goal is to determine effective principles of change in interventions for BFRBs. Therefore, assessing neurocognitive components using computer-based training programs can help identify the implicit processes underlying the disorder. The objective of the study is to examine the feasibility of using AAT to modify PSP action tendencies, and potentially improve PSP symptoms. The investigators predict that individuals with PSP will have a pathological approach tendency towards skin as measured by the Approach-Avoidance Assessment (AAA). Therefore, AAT will promote reduction of approach to skin stimuli. To retrain one's action tendencies the investigators will randomize participants to the following training conditions: Avoidance Training (AvT; avoidance of skin stimuli), Approach Training (ApT; approach skin stimuli), or Placebo Training (PT; equal approach/avoidance of skin stimuli). The investigators will also administer an eye-tracking task to assess visual gaze response to pictures of irregular skin and neutral stimuli to evaluate training-induced changes in action tendencies. Previous studies have shown the AAT's success in reducing action tendencies and symptoms in other addictions like problematic alcohol use and cigarette smoking Therefore, AAT may prove effective in modifying the behavioral addiction of PSP. Sixty adults with PSP will be randomly assigned to (a) approach training (b) avoidance training or (c) placebo training. All participants will then be sent a follow-up survey approximately two weeks after completion of the main study to determine changes in symptoms. This pilot study is expected to guide the development of an accessible, cost-efficient, and effective cognitive training programs for individuals with PSP.

ELIGIBILITY:
Inclusion Criteria:

1. A current diagnosis of skin picking
2. Moderate symptoms of skin picking a Skin Picking Severity Scale (SPS) score of ≥ 7
3. Ages 18-60,
4. Fluent English speakers.

Exclusion Criteria:

1. Self-reported visual impairment that cannot be adjusted and will prevent participants from clearly recognizing words and pictures on computer screen
2. A positive diagnosis of bipolar disorder or psychotic disorder

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2020-06-22 (Actual); Study Completion 2020-06-22 (Actual)

PRIMARY OUTCOMES:
Changes in Behavioral Approach Tendency After a Single Training Session | Pre-training, Post-training (30-minutes after training)
  This assessment evaluates behavioral approach (i.e., reaction time to avoid - reaction to approach) to irregular skin stimuli before and after training (i.e., the AAT). The investigators will measure reaction time to approach irregular skin stimuli before training and then measure changes in reaction time to approach irregular skin stimuli immediately after training (i.e., post-training; defined as 30 minutes after training). The investigators will then average the reaction time for each group, and then evaluate statistical differences between groups.

SECONDARY OUTCOMES:
Changes in Urges to Pick After Training | Pre-training, Post-training (30-minutes after training)
  Evaluates urges to pick before and immediately after training (same-day post-training), using a behavioral approach task. Urges will be rated on a scale of 0 to 100, where 0 indicates no urges to pick and 100 indicates severe urges to pick. Participants will rate urges to pick for a total of 3 minutes and identify different areas where they feel the urge to pick. The investigators will then average the differences in urges within groups, and then evaluate statistical differences between groups.
Changes in scores on the Skin Picking Scale-Revised (SPS-R). | Pre-training, 2 weeks (follow-up)
  This 8-item scale measures skin picking severity (4 items) and impairment (4 items). The scale ranges from 0 to 32, where higher scores represent worse skin picking severity. Sub-scales ranges from 0 to 16, where the scores are summed to compute a total score.

CONTACTS AND LOCATIONS:
Overall Officials: Han Joo Lee, Ph.D., Principal Investigator — University of Wisconsin, Milwaukee
Locations (1):
- Psychology Clinic, University of Wisconsin-Milwaukee, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No